CLINICAL TRIAL: NCT02439697
Title: A Cohort Study of Conversion From Aranesp® to NESP® for the Treatment of Anemia in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Mok Ming Yee, Resident Specialist, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.2 18thApril, 2015
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Anemia; End Stage Renal Failure on Dialysis
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Darbepoetin alfa (NESP®) same dose (Experimental): Patients on stable low dose Aranesp® (darbepoetin alfa manufactured by Amgen®) (on 20mcg preparations or on 40mcg every 2 weeks or less) will be converted to the same dose of NESP® (darbepoetin alfa manufactured by Kirin®)
  Interventions: Other: Darbepoetin alfa
- Extended dosing Darbepoetin alfa (NESP®) (Experimental): Patients on stable dose of Aranesp® (darbepoetin alfa manufactured by Amgen®) will be converted to higher dose preparation of NESP® (darbepoetin alfa manufactured by Kirin®) 40 or 120 mcg preparations) with extended dosing intervals. The total dose of Darbepoetin alpha remains the same.
  Interventions: Other: Darbepoetin alfa
- Darbepoetin alfa (NESP®) 120mcg (Experimental): Patients on Aranesp® 100 mcg preparation (darbepoetin alfa manufactured by Amgen®) will be switched to the NESP® (darbepoetin alfa manufactured by Kirin®)120mcg preparation with slight increase in dosing interval according to the conversion
  Interventions: Other: Darbepoetin alfa

INTERVENTIONS:
Other: Darbepoetin alfa — Conversion from Aranesp® to NESP®
  Other Names: NESP

SUMMARY:
This is a prospective single-arm open-labeled cohort study on dialysis patients of the conversion from Aranesp® to NESP® for the treatment of anemia. The primary outcome of the study is the haemoglobin level after conversion to NESP® after 6 months. Secondary outcomes include the variability in haemoglobin level, average weekly dose of erythropoietin, safety profile of NESP®, patients' subjective assessment of fatigue and injection pain after the conversion.

DETAILED DESCRIPTION:
Currently in Hong Kong, Aranesp®, manufactured by Amgen® is the only available Darbepoetin alpha licensed. NESP®, a Darbepoetin alpha agent manufactured by Kirin®, will be replacing Aranesp®.It is important to evaluate the therapeutic equivalence of the two agents, and its efficacy, tolerability and safety profile in the treatment of anemia in dialysis patients. Moreover, a new maximum preparation of NESP 120® microgram will be available to replace the Aranesp® 100 microgram prefilled syringe at the same cost. This larger Darbepoetin alpha preparation may allow extension of dosing intervals. This may subsequently allow cost saving and better convenience to medical staff and patients.

The objectives of this project are:

1. To investigate the effectiveness of NESP® in the achieving a stable anemia control in chronic dialysis patients with the same dose conversion from Aranesp®
2. To investigate the effectiveness of increasing the dosing interval of NESP® (but maintaining the same total dose) in sustaining a stable anemia control in chronic dialysis patients
3. To explore the possibility of cost saving in administering a larger dose NESP® but at an extended interval

   Patients will be divided into 3 groups.

   Group A. Same dose conversion group

   • Patients on stable low dose Aranesp® (on 20mcg preparations or on 40mcg every 2 weeks or less) will be converted to the same dose of NESP®

   Group B. Attempt extension of dosing interval with higher dose of NESP® preparations

   • Patients on stable dose of Aranesp® will be converted to higher dose preparation of NESP® (40 or 120 mcg preparations) with extended dosing intervals.

   Group C. Attempt dosage saving with 120 mcg preparation

   • Patients on Aranesp® 100mcg will be switched to the NESP® 120mcg preparation with slight increase in dosing interval

ELIGIBILITY:
Inclusion Criteria:

* Adult Chinese patients (age greater than or equal to 18)
* on long-term dialysis for at least 3 months
* on Aranesp® treatment for at least 3 months
* stable hemoglobin level within the range of 9 to12 g/dL, on the same stable dose of Aranesp® within the past 2 months.
* Minimum weekly kT/V of 1.7 for peritoneal dialysis patients and 1.2 per haemodialysis session for haemodialysis patients
* Able to give informed consent

Exclusion Criteria:

Presence of

* thalassaemia
* haematological diseases
* severe hyperparathyroidism (PTH >90 pmol/L)
* iron, vitamin B12 or folate deficiency
* uncontrolled malignancy
* active blood loss or hemolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Haemoglobin | 6 months

SECONDARY OUTCOMES:
Variability in haemoglobin level | 6 months
average weekly dose of erythropoietin | 6 months
safety profile of NESP | 6 months
  Blood pressure, Questionnaire on the occurrence of side-effects such as seizure, pure red cell aplasia, etc.
Subjective assessment of fatigue | 6 months
  Visual Analogue Fatigue Scale
Subjective assessment of pain | 6 months
  Numeric Pain Numeric Pain Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Ming Yee Mok, MBBS FHKAM, Principal Investigator — Queen Mary Hosptial, the University of Hong KOng; Tak Mao Chan, MBBS FRCP, Study Director — Queen Mary Hospital, the University of Hong Kong
Locations (1):
- Division of Nephrology, Department of Medicine, Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Vanrenterghem Y, Barany P, Mann JF, Kerr PG, Wilson J, Baker NF, Gray SJ; European/Australian NESP 970200 Study Group. Randomized trial of darbepoetin alfa for treatment of renal anemia at a reduced dose frequency compared with rHuEPO in dialysis patients. Kidney Int. 2002 Dec;62(6):2167-75. doi: 10.1046/j.1523-1755.2002.00657.x. PMID 12427142
- [Background] Galle JC, Claes K, Kiss I, Winearls CG, Herlitz H, Guerin A, Di Giulio S, Suranyi MG, Bridges I, Addison J, Farouk M. An observational cohort study of extended dosing (once every 2 weeks or once monthly) regimens with darbepoetin alfa in patients with chronic kidney disease not on dialysis: the EXTEND study. Nephrol Dial Transplant. 2012 Jun;27(6):2303-11. doi: 10.1093/ndt/gfr677. Epub 2011 Dec 2. PMID 22140136
- [Background] Hiramatsu M, Kubota M, Iwasaki M, Akizawa T, Koshikawa S; KRN321 A09 Study Group. Darbepoetin alfa (KRN321) administered intravenously once monthly maintains hemoglobin levels in peritoneal dialysis patients. Ther Apher Dial. 2008 Feb;12(1):19-27. doi: 10.1111/j.1744-9987.2007.00525.x. PMID 18257808
- [Background] Suzuki H, Inoue T, Watanabe Y, Kikuta T, Sato T, Tsuda M, Uchida K. Testing a single monthly dose of darbepoetin alpha to maintain hemoglobin levels in continuous ambulatory peritoneal dialysis patients. Adv Perit Dial. 2011;27:60-4. PMID 22073831